CLINICAL TRIAL: NCT05065255
Title: Study of the Criteria for Choosing Speedicath Catheters During the Initiation of Self-catheterization
Acronym: Eva
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laboratoires Coloplast S.A.S (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A00579-32
Record Dates: First submitted 2021-08-10; First posted 2021-10-04 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Adult subjects with neurogenic or non-neurogenic urinary tract disorders, newly initiated to ASI, and users of the SpeediCath line of catheters.
  Interventions: Device: SpeediCath® catheters

INTERVENTIONS:
Device: SpeediCath® catheters — Patients using SC catheters will be followed up in order to understand the major criteria in the choice of the catheter by the patients.

SUMMARY:
To date, there is no objective data to help in the choice of the type of catheter to offer to the patient according to his or her needs. Although it is now known that the quality of life of patients practicing intermittent self catheterisation is dependent on multiple factors, there is little data on the factors that facilitate or hinder adherence to intermittent self catheterisation during the first six months after initiation of intermittent self catheterisation. The prospective multicenter exploratory observational study that the sponsor wishes to conduct aims to determine what criteria preside over patient choice of SpeedyCath (SC) leads. This information would allow us to set up a personalized advice with each patient in the future, with the aim of proposing the SC catheter best adapted to his needs. The study population will consist of adults with neurogenic or non-neurogenic urinary disorders that warrant the use of intermittent self catheterisation, with intermittent self catheterisation education occurring at the time of inclusion. Patients should be autonomous in the practice of intermittent self catheterisation, and the minimum expected duration of follow-up should be greater than or equal to 6 months. Only patients who choose to use SpeediCath leads will be included in the study.

DETAILED DESCRIPTION:
Urinary self-catheterization consists of emptying the bladder oneself by inserting a catheter into the urethra. It is the reference method in case of dysfunctions of the bladder emptying phase, in particular in case of complete urinary retention or complete or incomplete bladder emptying with sub bladder obstruction. Neurological pathologies such as spinal cord injury, multiple sclerosis, multisystematic atrophy, peripheral neuropathies, Parkinson's disease, and stroke, may be the cause of bladder disturbances. These disturbances may also be caused by pelvic denervations as a result of enlarged pelvic surgeries or radiotherapy for the treatment of gynecological, urological or digestive cancers.

The objective of the implementation of intermittent self-catheterization (ISC) is to reduce the morbidity related to bladder and bowel dysfunction and to improve the quality of life of patients by making them more autonomous.

It involves a rigorous learning phase for the patient and a phase of acceptance of this new mictional mode.

When ISC is indicated, training is provided to the patient to enable him/her to manage daily catheterization. The objectives of this training are to understand, perform, monitor and adapt self-care. This training, mainly provided by the nursing staff and/or a specialist physician, is usually provided during a hospitalization. After returning home, the patient continues to be monitored by the specialist physician and the nursing team to evaluate the mastery of the technique (possibly reviewing the gesture and ensuring the adequacy of the catheter), the patient's adaptation to the practice of ISC, his compliance with the associated rules (frequency and regularity of catheterization, volume of urine) and any complications. A first visit is usually made between 3 and 12 weeks, then a second one after 6 months of use.

However, this therapeutic patient education (TPE), even when carried out by trained personnel, is not necessarily sufficient for immediate acceptance and adherence to self-catheterization in the medium to long term.

It is important that the patient is involved in his or her choice of equipment, since the decision to self-catheterize is usually made by the physician, and that the benefits of self-catheterization outweigh the constraints. The patient must be guided and involved in the choice of catheter during this learning phase, which will ensure better compliance and future adherence to treatment.

The interest of this study is therefore to better understand the real motivations of the patient in the choice of the catheter. This will undoubtedly make it possible to improve either the equipment itself or certain FTE sequences in the future by insisting on the problematic or questioning points in terms of the choice of catheter proposed to the patient by the caregiver. The determinants of the patient's choice are all the more important as there are a very large number of catheters on the market.

Coloplast offers the SpeediCath® (SC) range of ready-to-use self-lubricating hydrophilic catheters. This range is designed to cover the different needs of patients, providing them with probes of different length, flexibility, shape and ergonomics. There are 3 types of catheters adapted to women (SC Standard®, SC Compact® and SC Compact Set, SC Compact Eve®), and 3 types of catheters adapted to men (SC Standard®, SC Compact® and SC Compact Set, SC Flex®).

Concerning the technical specificities, a systematic review of the literature concluded that hydrophilic catheters (with a lubricant attached to the catheter) provide a benefit in terms of safety and quality of life, particularly in patients with spinal cord injuries. SC® catheters significantly reduce trauma to the urinary tract by reducing friction. Another study also showed that SpeediCath catheters were significantly faster, more convenient, and more discreet to use than a non-ready-to-use hydrophilic catheter (need to activate lubricant). The superiority of SpeediCath Compact Male and Female catheters in terms of quality of life compared to reference catheters was demonstrated in a randomized study using the specific validated ISC-Q questionnaire and has been retained and valued by the CNEDiMTS

To date, there is no objective data to help in the choice of the type of catheter to propose to the patient according to his needs. Although it is now known that the quality of life of patients using ISC is dependent on multiple factors, there is little data on the factors that facilitate or hinder adherence to ISC during the first six months after initiation of ISC. The prospective multicenter exploratory observational study that the sponsor wishes to conduct aims to determine the criteria that govern patient choice of SC leads. This information would allow us to set up a personalized advice with each patient in the future, with the aim of proposing the SC catheter best adapted to his needs. The study population will consist of adults with neurogenic or non-neurogenic urinary disorders that warrant the use of ISC, with ISC education occurring at the time of inclusion. Patients should be autonomous in the practice of ISC, and the minimum expected duration of follow-up should be greater than or equal to 6 months. Only patients who have chosen to use SpeediCath leads will be included in the study.

Numerous criteria will be collected to allow a detailed analysis of the modalities of choice of the type of SC probe. This collection involves the use of self-questionnaires for the patients. These questionnaires will be collected during the usual follow-up of the patient, including a visit at the time of the ASI education, a follow-up visit around 3 to 12 weeks (depending on the practices of the investigating center) and a second follow-up visit around 6 months.

Acceptance of ISC will be measured by the Intermittent Catheterization Acceptance Test (I-CAT). This is a patient questionnaire developed by the Groupe d'Études de Neuro-Urologie de Langue Française (GENULF) and validated in French in 2016 during a prospective multicenter study of 201 neurological and non-neurological patients. The I-CAT allows for a better assessment and understanding of the psychological barriers encountered by patients in relation to ISC. The questionnaire consists of 14 questions, with a minimum score of 0 for perfect acceptance and a maximum score of 56 characterizing the least possible acceptance.

The difficulties encountered by patients during ASI will be measured by the "Intermittent Catheterization Difficulty Questionnaire" IC-Di-Q. This is a patient questionnaire validated in French, and its purpose is to evaluate the difficulties encountered during the performance of ISA. In 13 questions, it explores numerous factors such as pain, blockage, bleeding, spasticity, and urethral sphincter spasm, in terms of frequency of occurrence and intensity. The purpose of this questionnaire is to identify the difficulties encountered by patients, and to monitor their evolution after the implementation of alternatives or solutions (including the adaptation of the type of catheter).

Patient adherence to ISC will be measured by the Intermittent Catheterization Adherence Scale (I-CAS). This is a patient questionnaire validated in French with 8 questions, 7 of which have a binary answer (yes/no), and one with 5 suggested answers. The score ranges from 0 for strong adherence to ISC to 8 for very weak adherence.

A study-specific self-questionnaire was also created with the support of the Scientific Advisory Board to determine the reasons for the patient's choice of catheter. This questionnaire includes criteria independent of the patient (e.g. advice from the nurse), and criteria specific to the patient (e.g. ease of use, discretion).

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 years of age or older
* Subject having been informed of the study and having decided to participate (no opposition)
* Subject affiliated to a social security system or entitled to it
* Subject with neurogenic or non-neurogenic urinary disorders, justifying the use of the ISC to empty the bladder
* Subjects who have received their first ISC education at the time of inclusion
* Subject with an expected duration of ISC of at least 6 months
* Subject has been presented with at least two types of SC catheters and has chosen to use the SpeediCath line of catheters as their first self-catheterization catheter
* Able to perform ISC independently
* Subjects who have been recommended by their healthcare professional to perform catheterization at least 4 times per day

Exclusion Criteria:

* Vulnerable subject according to the regulations in force
* Pregnant, parturient or nursing woman;
* Subject deprived of liberty by judicial, medical or administrative decision;
* Minor subject ;
* Subject protected by law or unable to give consent
* Subject who is not affiliated or not a beneficiary of a social security system;
* Subject falling into several of the above categories;
* Subject who has refused to participate in the study
* Subject participating in an interventional clinical study
* Subjects who, in the opinion of the investigator, have cognitive problems that prevent them from answering a questionnaire or for whom assessment could be problematic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to all adult subjects with neurogenic or non-neurogenic urinary disorders, newly initiated to ISC, and using the SpeediCath line of catheters.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire for the choice of the catheter | At visit 3 : 6 months
  A study-specific self-administered questionnaire was created with the support of the Scientific Advisory Board to determine the reasons for the patient's choice of catheter. This questionnaire contains 18 questions, including criteria independent of the patient (e.g. advice from the nurse), and criteria specific to the patient (e.g. ease of use, discretion).

SECONDARY OUTCOMES:
Patient questionnaire for the choice of the catheter | At baseline
  A study-specific self-administered questionnaire was created with the support of the Scientific Advisory Board to determine the reasons for the patient's choice of catheter. This questionnaire contains 18 questions, including criteria independent of the patient (e.g. advice from the nurse), and criteria specific to the patient (e.g. ease of use, discretion).
Patient satisfaction | At visit 2 : 3 to 12 weeks
  Determined by a 0 to 5 points visual analog scale, 0 is the worst possible satisfaction, and 5 is the best possible satisfaction
Patient satisfaction | At visit 3 : 6 months
  Determined by a 0 to 5 points visual analog scale, 0 is the worst possible satisfaction, and 5 is the best possible satisfaction
"Intermittent Catheterization Difficulty Questionnaire" IC-Di-Q | At visit 2 : 3 to 12 weeks
  This is a patient questionnaire validated in French.The purpose of this questionnaire is to identify the difficulties encountered by the patients and to follow their evolution after the implementation of alternatives or solutions (including the adaptation of the type of catheter). In 13 questions, it explores numerous factors such as pain, blockage, bleeding, spasticity, and urethral sphincter spasm, in terms of frequency of occurrence and intensity.
"Intermittent Catheterization Difficulty Questionnaire" IC-Di-Q | At visit 3 : 6 months
  This is a patient questionnaire validated in French.The purpose of this questionnaire is to identify the difficulties encountered by the patients and to follow their evolution after the implementation of alternatives or solutions (including the adaptation of the type of catheter). In 13 questions, it explores numerous factors such as pain, blockage, bleeding, spasticity, and urethral sphincter spasm, in terms of frequency of occurrence and intensity.
Catheterization Adherence Scale (I-CAS) | At visit 2 : 3 to 12 weeks
  This is a patient questionnaire validated in French with 8 questions, 7 of which have a binary response (yes/no), and one with 5 suggested answers. The score ranges from 0 for strong adherence to ASI to 8 for very weak adherence.
Catheterization Adherence Scale (I-CAS) | At visit 3 : 6 months
  This is a patient questionnaire validated in French with 8 questions, 7 of which have a binary response (yes/no), and one with 5 suggested answers. The score ranges from 0 for strong adherence to ASI to 8 for very weak adherence.
Intermittent Catheterization Acceptance Test (I-CAT) questionnaire | At baseline
  The I-CAT allows for a better assessment and understanding of the psychological barriers encountered by patients in relation to ISA. The questionnaire consists of 14 questions, with a minimum score of 0 for perfect acceptance and a maximum score of 56 characterizing the least possible acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard AMARENCO, Pr., MD, Principal Investigator — Hôpital Tenon
Locations (37):
- France (37):
  - Centre hospitalier d'Aulnay sous bois, Aulnay-sous-Bois
  - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre auterive, Auterive
  - Centre Calvé- Fondation Hopale, Berck
  - Tour de Gassies, Bruges
  - CHU de Caen, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre médical Germaine Revel, Chamalières
  - Hôpitaux civil de Colmar, Colmar
  - CHU Le Bocage, Dijon
  - Hôpital Raymond Poincaré, Garches
  - Centre Hospitalier de Gonesse, Gonesse
  - CHU GrenobleAlpes, La Tronche
  - Hôpital Swynghedauw, Lille
  - CHU Limoges, Limoges
  - Clinique Saint Martin, Marseille
  - CHU de Timonnes, Marsillargues
  - Hôpital Lapeyronie, Montpellier
  - Institut Mutualiste Montpelliérain- Beau soleil, Montpellier
  - CHU de Nancy, Nancy
  - Hôpital Saint jacques, Nantes
  - Hôpital Pasteur 2 - CHU de Nice, Nice
  - Hôpital Tenon, Paris
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Centre PSR, Perpignan
  - CMMRF Kerpape, Ploemeur
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - Hôpital Victor Provo, Roubaix
  - CHU Rouen, Rouen
  - Hopital Charles Nicolle, Rouen
  - Hôpital Bellevue, CHU de SAINT ETIENNE, Saint-Etienne
  - Hôpital Henry Gabrielle, Saint-Genis-Laval
  - Centre de l'Arche, Saint-Saturnin
  - Nouvel Hôpital Civil, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT05065255/Prot_000.pdf